CLINICAL TRIAL: NCT06894056
Title: "Cerrahi Eksizyon ve Greft Ile Tedavi Edilmiş Olan Nonmelanoma Deri Kanseri Hastalarda Greft Donör Alanı Ile Post Operatif 3. Ayda Yaşam Kalitesinin İlişkisinin Araştırılması"
Brief Title: Investigating the Effects of Orienting Skin Grafts Parallel to Skin Tension Lines on Quality of Life in Head and Neck Located Basal Cell Carcinoma
Status: Completed | Type: Observational
Sponsor: Sifa Okulu - Independent Research Center of Dermatology and Venereology (Other)
Responsible Party: Principal Investigator, Hilayda Karakok Kısla, Principal Investigator, Sifa Okulu - Independent Research Center of Dermatology and Venereology
Other Study IDs: KAEK258
Record Dates: First submitted 2025-03-17; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Basal Cell Cancer; Grafting
Keywords: basal cell carcinoma; skin tension lines; grafting; cosmetic outcome; quality of life
MeSH Terms: conditions — Neoplasms, Basal Cell; Carcinoma, Basal Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Control patients were selected either from patients with head and neck located BCC's who were treated with excision with grafting harvested from clavicular region with no specific attention in terms of orientation of skin tension lines
- Group 2: Group two was selected from patients with BCC located at head and neck and who underwent a grafting method. A skin tension lines oriented approach was applied and grafts were harvested from a color matched cosmetic area in these patients.

SUMMARY:
The goal of this observational study is to learn about the effect of orienting graft for treatment of skin cancer in patients who undergo skin cancer excision and grafting for their skin cancer. The main question to answer is

Does orienting the grafts parallel with skin tension lines have any effect on quality of life or cosmetic results?

Participants who already underwent or planned to undergo an excision and grafting procedure will answer a qaulity of life tool and cosmetic results will be evaluated by two seperate dermatologist.

ELIGIBILITY:
Inclusion Criteria:

* Patients with nodular basal cell carcinomas with a tumor size equal or less than 12 millimeters
* A history of surgical excision and grafting

Exclusion Criteria:

* Immunosuppressed patients
* Recurrent tumors
* Patients with BCC's that arose from the previously irradiated area
* Gorlin's Syndrome diagnosis
* Illiterate individuals
* İmpaired cognitive functions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants were selected from the individuals who were admitted or referred to study center (Dr. Hilayda Karakok Private Practice of Dermatology and Venereology).
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2021-11-20 (Actual); Primary Completion 2025-02-22 (Actual); Study Completion 2025-02-22 (Actual)

PRIMARY OUTCOMES:
Quality of Life Outcome | At least three months after surgery and grafting
  Quality of life outcome was measured by the disease specific tool "Skin Cancer Quality of Life Impact Tool", SCQOLIT is a 10 item questionnaire and each item has 4 answers, total score is ranged between 0-30. Higher scores mean worse outcomes.
Quality of Life - General | At least three months after surgery and grafting
  Dermatology Quality of Life Index was also used to evaluate quality of life as a general quality of life tool. DLQI is alsa a ten item tool with a total score range between 0-30. Higher scores mean worse outcomes.

SECONDARY OUTCOMES:
Cosmetic Outcome | At least three months after the surgery and grafting
  Cosmetic outcome of the grafting at the third month, evaluated by two different dermatologists one of whom did the operations. As the initial part of the study was during pandemic precautional period second surgeon the results via photographs (teleconsultation). Visual analog scala is used, the scale is ranged between 0-8, higher scores meaning better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Hilayda Karakök Kışla, MD, Specialist of Dermatology, Principal Investigator — Dr. Hilayda Karakök Muayenehanesi
Locations (1):
- Dr. Hilayda Karakök Deri ve Zührevi Hastalıklar Muayenehanesi, Ordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Due to the sensitivity of the personal information contained within the research data, for the confidentiality and privacy of our participants our team has not yet decided upon sharing. Consequently, while an anonymized version of the data might be shared, individual participant data will not be disclosed to protect their identity and personal information. This approach ensures compliance with ethical standards and regulations related to data privacy.